CLINICAL TRIAL: NCT02532166
Title: Incidence of Esophageal Lichen Planus in Patients With Known Oral Lichen Planus. Diagnostic Value of White Light Endoscopy, Narrow Band Imaging and Chromoendoscopy for Detection of Esophageal Manifestation in Patients With Oral Lichen.
Brief Title: Incidence of Esophageal Lichen Planus in Patients With Known Oral Lichen Planus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Andrea Riphaus, PD Dr. Andrea Riphaus, Ruhr University of Bochum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-4072
Record Dates: First submitted 2015-08-17; First posted 2015-08-25 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Lichen Planus
Keywords: narrow band imaging; Chromoendoscopy; Lugol
MeSH Terms: conditions — Lichen Planus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Esophageal lichen planus (Other): White light endoscopy compared to narrow band imaging and chromoendoscopy with Lugol for detection of esophageal lichen.
  Interventions: Other: Esophageal lichen planus

INTERVENTIONS:
Other: Esophageal lichen planus — White light endoscopy compared to narrow band imaging and Lugol for detection of esophageal lichen.

SUMMARY:
The lichen planus is a mucocutaneous disease of unknown etiology with an incidence of 1-2%, that affects in 30-70% of cases either the mucosa of the mouth, or partly in combination with infection of the skin, the oral with his known premalignant potential in up to 2-3% predisposed to the development of an oral squamous cell carcinoma.In rare cases, there is also an manifestation of the lining of the esophagus, which can then be associated with symptomatic strictures of the esophagus.

The value of moreover increasingly established endoscopic imaging procedures are investigated as well as data of the natural long-term outcome in esophageal lichen planus infestation especially in view of malignant transformation.

DETAILED DESCRIPTION:
The lichen planus is a mucocutaneous disease of unknown etiology that manifests itself with an incidence of 1-2% in 30-70% of cases either at the mucosa of the mouth, or partly in combination with infection of the skin, the oral with his known premalignant potential in up to 2-3% predisposed to the development of an oral squamous cell carcinoma. In rare cases, there is also an manifestation of the lining of the esophagus, which can then be associated with symptomatic strictures of the esophagus. In addition, four cases have been reported with esophageal squamous cell carcinoma in patients with esophageal lichen planus.

The value of moreover increasingly established use of narrow-band imaging (a process for improving the detection of early cancers in the gastrointestinal tract by creating a maximum contrast between outright and altered mucosa, which could have already shown an improved detection rate of early lesions of the esophagus as well as squamous cell carcinoma), or the chromoendoscopy has means for example Lugol solution in correlation to the histopathologic findings in lichen planus), has not been investigated to date.

Also, data of the natural long-term outcome in esophageal lichen planus infestation especially in view of malignant transformation are currently not available.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Known lichen planus of the oral mucosa

Exclusion Criteria:

* Severe cardiopulmonary disease - ASA (American Society of Anaesthesiology) class > III
* Antisecretory and nonsteroidal anti-inflammatory medication within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Value of additional endoscopic enhancing imaging methods for detection of esophageal lichen planus. | 3-5 years

SECONDARY OUTCOMES:
Natural long-term incidence of esophageal lichen planus in patients with known oral lichen. | 3-5

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Riphaus, PD Dr, Principal Investigator — Department of Medicine, KRH Laatzen
Locations (2):
- Germany (2):
  - Department of Medicine, Bochum
  - Klinikum Agness Karll Laatzen, Laatzen

REFERENCES:
- [Background] Quispel R, van Boxel OS, Schipper ME, Sigurdsson V, Canninga-van Dijk MR, Kerckhoffs A, Smout AJ, Samsom M, Schwartz MP. High prevalence of esophageal involvement in lichen planus: a study using magnification chromoendoscopy. Endoscopy. 2009 Mar;41(3):187-93. doi: 10.1055/s-0028-1119590. Epub 2009 Mar 11. PMID 19280529